CLINICAL TRIAL: NCT04944095
Title: Serology Testing (Antibody Levels) With Time Following SARS-CoV-2 (Covid-19) Vaccinations in Residents of Nursing, Extended Care, and Over-55 Communities
Brief Title: Change in Antibody Levels Following SARS-CoV-2 (Covid-19) Vaccinations
Acronym: Covid-19-Abs
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Dr. Sidney J. Stohs (Other)
Collaborators: Telos Healthcare, LLC (Unknown); Remarkable Healthcare (Unknown); The Alden Network (Unknown); Churchill Residential (Unknown); Corridor Mobile Medical Services (Unknown); Siemens Healthineers USA (Unknown); HealthTrackRX/AIT (Unknown); Abri Healthcare Services, LLC (Unknown); Brookdale Senior Living, Inc. (Unknown); Cantex Healthcare Centers, LLC (Unknown); Christian Care Centers, Inc. (Unknown); Cottonwood Creek Healthcare Community (Unknown); Creative Solutions in Healthcare, Inc. (Unknown); Dynasty Healthcare LLC (Unknown); Midlothian Care Center (Unknown); Nexion Health, Inc. (Unknown); Optimum Healthcare, Inc. (Unknown); Paramount Healthcare Consultants, LLC (Unknown); Priority Healthcare, Inc. (Unknown); Revelations Healthcare Group, LLC (Unknown); Southwest Long Term Care, LLC (Unknown); Stonegate Senior Living, LLC (Unknown); Summit Healthcare, Inc. (Unknown); TGR Healthcare, LLC (Unknown); Trinity Healthcare, LLC (Unknown)
Responsible Party: Sponsor-Investigator, Dr. Sidney J. Stohs, EVP Global Scientific Affairs, Boston Biopharm, Inc.
Organization: Boston Biopharm, Inc. (Other)
Other Study IDs: SARS-CoV-2 Antibodies Levels
Record Dates: First submitted 2021-06-24; First posted 2021-06-29 (Actual); Last update posted 2022-08-29 (Actual); Status verified 2022-08

CONDITIONS: Covid-19; Subjects Vaccinated Against Covid-19
Keywords: IgG antibodies; total antibodies (IgG+ IgM); age 55 and above; post-covid-19 vaccination; Confounding factors
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: None Retained — Blood samples will be drawn from an appropriate vein as the median cubital vein. Blood samples of 3.0 ml will be collected in mind green-topped plastic, BD Vacutainer PST blood collection tubes containing lithium-heparin using 21-23 gage needles, and stored at room temperature for not more than 6 hours before centrifugation on site to prepare plasma which will be sent to the analytical laboratory. The blood samples will be packed in biohazard, plastic leak-proof bags, and transported in insulated containers with cold packs to ensure the integrity of the samples, as necessary. Plasma samples will be stored at 2-8°C if not tested within 8 hours, and frozen if not tested within 14 days.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- SARS-CoV-2 Antibody Levels: This is a single arm study by Southlake Diagnostics Inc. whereby changes in plasma antibody levels (IgG and total) are determined over 12 months on individuals residing in over 300 associated nursing homes, extended care facilities and over-55 residences following vaccination with one of the authorized SARS-CoV-2 vaccines (Pfizer, Moderna or J &J). No interventions are involved. The investigators are not responsible for administering the vaccines or determining subject eligibility or willingness to receive the vaccine. Blood samples will be drawn and plasma IgG and total antibodies will be determined at baseline, 3, 6, 9 and 12 months post-vaccination.
  Interventions: Other: Change in SARS-CoV-2 Antibody Levels

INTERVENTIONS:
Other: Change in SARS-CoV-2 Antibody Levels — Changes in plasma antibody levels over 12 months will be determine post-vaccination with one of the authorized SARS-CoV-2 vaccines.
  Other Names: No other names apply

SUMMARY:
Limited information is available regarding the effects of various factors that may influence the duration and effectiveness of severe acute respiratory syndrome coronavirus 2 (SARS CoV-2) vaccinations. This virus causes Covid-19. Such factors include age, disease states, general immunocompetence, and use of various drugs. The results of this study by Southlake Diagnostics Inc. will provide base-line antibody (IgG and total) data regarding the extent to which the results from this test can be interpreted as an indication or degree of protection from infection after vaccination with one of the three authorized SARS-CoV-2 vaccines (Pfizer, Moderna or J& J), with information regarding various confounding factors. The study will include 30,000 male and female or more residents associated with over 300 nursing homes, extended care facilities and over-55 communities as well as staff associated with these facilities. Demographic data of the subjects including characteristics, and medical histories including concomitant medications and disease states/conditions will be collected and submitted to Southlake Diagnostics for analysis via the REDCap platform (described below). Various possible statistical correlations will be assessed.

DETAILED DESCRIPTION:
Subjects:

This study protocol will be registered with ClinicalTrails.gov and approval by an independent ethics committee. All subjects will be provided detailed written information concerning the trial, and will be required to give written consent to participate in the study. The investigators will collect blood samples from residents associated with over 300 nursing homes, extended care facilities and over-55 communities which have agreed to participate in the study at baseline (when available), and at 3, 6, 9 and 12 month timepoints post-vaccination with one of the three authorized SARS-CoV-2 vaccines. The plasma samples will be analyzed by Southlake Diagnostics.

The study will include up to 10,000 male and female residents of nursing homes, extended care facilities and over-55 communities as well as staff associated with these facilities. Demographic data of the subjects including characteristics, and medical histories including concomitant medications and disease states/conditions will be collected.

Blood Sample Collection:

A standard operating procedure (SOP) has been developed by Southlake Diagnostics to establish a standardized procedure for establishing a safe and appropriate location and method for obtaining human blood samples. This SOP incorporates regulations and recommendations from the Occupational Safety and Health Administration (OSHA) Needlestick Safety and Prevention Act (29 CFR 1910.1030). Blood draws conducted by Southlake Diagnostics personnel will abide by this SOP.

The OSHA Bloodborne Pathogen Standard, (29 CFR 1910.1030) defines the required usage of Safety Engineered Sharps Devices for any clinical research (including blood draws and injections). All personnel conducting human blood draws are required to use Safety Engineered Sharps Devices.

Personnel conducting blood draws are required to wear the appropriate personal protective equipment (PPE). The Clinical Operations team is responsible for verifying that laboratory personnel performing blood draws have appropriate training and experience in conducting human blood sampling.

Blood samples will be drawn from an appropriate vein as the median cubital vein. Blood samples of 3.0 ml will be collected in BD Vacutainer blood collection tubes containing lithium-heparin using 21-23 gage needles. The blood samples will be packed in biohazard, plastic leak-proof bags, and transported in insulated containers with cold packs to ensure the integrity of the samples, as necessary. Plasma will be prepared by centrifugation. Plasma samples will be stored at 2-8°C if not tested within 8 hours, and frozen if not tested within 14 days.

Analytical Methods:

IgG antibodies to SARS-CoV-2 in human plasma (lithium-heparin) will be determined using the Siemen's Atellica® IM SARS-CoV-2 IgG (sCOVG) assay (EUA Number: EUA202669) which is a chemiluminescent immunoassay intended for qualitative and semi-quantitative detection of IgG antibodies using the Atellica® IM Analyzer [1]. This SARS-CoV-2 IgG assay specifically detects IgG antibodies to the S1 receptor binding domain (RBD) antigen. IgG antibodies to SARS-CoV-2 are generally detectable in blood several days after initial infection or vaccination. The duration of time antibodies is present post-vaccination is not well characterized. The test will give an indication of the level of immunity that is provided by a vaccine for the SARS-CoV-2 virus which causes COVID-19.

The Atellica IM sCOVG assay is a fully automated 2 step sandwich immunoassay using indirect chemiluminescent technology. A direct relationship exists between the amount of SARS-CoV-2 IgG antibody present in a patient plasma sample and the amount of relative chemiluminescent light units (RLUs) detected by the system. Preparing master curves and performing calibrations of the system will be performed according to manufacturing instructions.

Results of the IgG antibody test are expressed as index values with an analytical measuring interval of 0.50-150.00 Index units. Plasma samples with index values >150 will be diluted and retested. Index values <1.00 will be considered negative (non-reactive) while values >1.00 will be considered positive (reactive) [1].

Total (IgM + IgG) antibodies to SARS-CoV-2 in human plasma (lithium-heparin) will be determined using the Siemen's Atellica® IM SARS-CoV-2 Total (COV2T) assay which is a chemiluminescent immunoassay intended for qualitative detection of total antibodies using the using the Atellica® IM Analyzer[1].

The Atellica IM COV2T assay is an automated immunoassay using indirect chemiluminescent technology [1]. Results of the total (IgM + IgG) antibody test are expressed as index values with an analytical measuring interval of 0.05-10.00 Index units. Index values <1.00 will be considered negative (non-reactive) while values >1.00 will be considered positive (reactive) [1]

[1]. https://www.siemens-healthineers.com/en-us/laboratory-diagnostics/assays-by-diseases-conditions/infectious-disease-assays/sars-cov-2-igg-assay

Data Management:

Demographic data of the subjects including characteristics, and medical histories including concomitant medications and disease states/conditions will be provided for each subject by the respective residence and inputted into the REDCap cloud platform (described below) by data input specialists employed by Southlake Diagnostics. Data entry will be checked by a second specialist for accuracy of entry. Standardized and approved terminology will be used for all entry parameters as height, weight, age, drug names, and disease states to ensure consistency of data entry. Data entry will be reviewed for accuracy of entry and validation by the Co-Principal Investigator (Dr. Robert Newton) who is responsible for this function, and the Principal Investigator.

Statistical Methods:

The laboratory will provide the certified statistician with a spread sheet of the data which will be sorted and analyzed as a whole and according to various parameters as gender, age groups, known disease states and immunocompetencies, physical characteristics and time after vaccination using a REDCap Cloud platform (www.redcapcloud.com/). This platform is advanced, compliant software for the management of all types of data associated with clinical studies. The system is Medical Dictionary for Regulatory Activities (MEdDRA) terminology certified, Clinical Data Interchange Standards Consortium (CDISC) compliant, and International Standards Organization (ISO) 27001 certified. The data will be sorted and analyzed for statistical significance and trends using various computer programs associated with the platform.

Information regarding overall duration and rate of decline of antibody levels as a function of time post-vaccination as well as the effects of confounding factors on antibody levels as a function of time will be determined. Information regarding antibody levels (IgG and total) and Covid-19 infection or reinfection, and approximate time at which a booster shot may be required will also be obtained relative to antibody levels. The large number of subjects in the overall study should enable statistical associations to be made between antibody levels and various potentially confounding and influencing factors. The data will be reviewed by the Principal Investigator and Co-PIs.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects of age 55 and above
* Has given voluntary, written, informed consent to participate in the study

Exclusion Criteria:

* Individuals who are unable to give informed consent.

Min Age: 55 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Residents and staff associated with nursing homes, extended care facilities and over-55 communities
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2021-08-10 (Actual); Primary Completion 2024-08-09 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in Plasma Antibody Levels with Time Following SARS-CoV-2 Vaccinations | Changes determined over 12 months (at baseline, 3,6, 9 and 12 months)
  Determination of plasma IgG and total (IgG + IgM) antibody levels with time

SECONDARY OUTCOMES:
Plasma Antibody Levels and Confounding Factors | Factors affecting changes over 12 months (determinations at baseline, 3,6, 9 and 12 months)
  A determination of whether factors as age, known immunocompetence, use of specific drugs, and specific disease states impact changes in plasma antibody levels over the 12 months of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Harry G Preuss, MD, Study Director — Georgetown University, washington, DC; Robert U Newton, Ph.D., Study Director — Edith Cowan University, Perth Western Australia
Locations (1):
- Southlake Diagnostics, Inc., Southlake, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
A plan is being developed whereby all IPD that is involved in publications will be shared with other investigators.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data regarding results associated with each of the three authorized vaccines will be shared upon completion of the study with other investigators and with their respective manufacturers. If the investigators determine that significant interim results may be of value and contribute to overall healthcare, for example to determine potential timing of booster vaccinations, this information will be made available to appropriate parties prior to publication.
Access Criteria: Governmental agencies as the Center for Disease Control, vaccine manufacturers, investigators with a track record in this area, and investigators with background deemed appropriate by the Principal and Co-Principal Investigators.

REFERENCES:
- [Background] VanBlargan LA, Goo L, Pierson TC. Deconstructing the Antiviral Neutralizing-Antibody Response: Implications for Vaccine Development and Immunity. Microbiol Mol Biol Rev. 2016 Oct 26;80(4):989-1010. doi: 10.1128/MMBR.00024-15. Print 2016 Dec. PMID 27784796
- [Background] Piccoli L, Park YJ, Tortorici MA, Czudnochowski N, Walls AC, Beltramello M, Silacci-Fregni C, Pinto D, Rosen LE, Bowen JE, Acton OJ, Jaconi S, Guarino B, Minola A, Zatta F, Sprugasci N, Bassi J, Peter A, De Marco A, Nix JC, Mele F, Jovic S, Rodriguez BF, Gupta SV, Jin F, Piumatti G, Lo Presti G, Pellanda AF, Biggiogero M, Tarkowski M, Pizzuto MS, Cameroni E, Havenar-Daughton C, Smithey M, Hong D, Lepori V, Albanese E, Ceschi A, Bernasconi E, Elzi L, Ferrari P, Garzoni C, Riva A, Snell G, Sallusto F, Fink K, Virgin HW, Lanzavecchia A, Corti D, Veesler D. Mapping Neutralizing and Immunodominant Sites on the SARS-CoV-2 Spike Receptor-Binding Domain by Structure-Guided High-Resolution Serology. Cell. 2020 Nov 12;183(4):1024-1042.e21. doi: 10.1016/j.cell.2020.09.037. Epub 2020 Sep 16. PMID 32991844
- [Background] Premkumar L, Segovia-Chumbez B, Jadi R, Martinez DR, Raut R, Markmann A, Cornaby C, Bartelt L, Weiss S, Park Y, Edwards CE, Weimer E, Scherer EM, Rouphael N, Edupuganti S, Weiskopf D, Tse LV, Hou YJ, Margolis D, Sette A, Collins MH, Schmitz J, Baric RS, de Silva AM. The receptor binding domain of the viral spike protein is an immunodominant and highly specific target of antibodies in SARS-CoV-2 patients. Sci Immunol. 2020 Jun 11;5(48):eabc8413. doi: 10.1126/sciimmunol.abc8413. PMID 32527802
- [Background] Wang H, Zhang Y, Huang B, Deng W, Quan Y, Wang W, Xu W, Zhao Y, Li N, Zhang J, Liang H, Bao L, Xu Y, Ding L, Zhou W, Gao H, Liu J, Niu P, Zhao L, Zhen W, Fu H, Yu S, Zhang Z, Xu G, Li C, Lou Z, Xu M, Qin C, Wu G, Gao GF, Tan W, Yang X. Development of an Inactivated Vaccine Candidate, BBIBP-CorV, with Potent Protection against SARS-CoV-2. Cell. 2020 Aug 6;182(3):713-721.e9. doi: 10.1016/j.cell.2020.06.008. Epub 2020 Jun 6. PMID 32778225
- [Background] Addetia A, Crawford KHD, Dingens A, Zhu H, Roychoudhury P, Huang ML, Jerome KR, Bloom JD, Greninger AL. Neutralizing Antibodies Correlate with Protection from SARS-CoV-2 in Humans during a Fishery Vessel Outbreak with a High Attack Rate. J Clin Microbiol. 2020 Oct 21;58(11):e02107-20. doi: 10.1128/JCM.02107-20. Print 2020 Oct 21. PMID 32826322
- [Background] Corbett KS, Flynn B, Foulds KE, Francica JR, Boyoglu-Barnum S, Werner AP, Flach B, O'Connell S, Bock KW, Minai M, Nagata BM, Andersen H, Martinez DR, Noe AT, Douek N, Donaldson MM, Nji NN, Alvarado GS, Edwards DK, Flebbe DR, Lamb E, Doria-Rose NA, Lin BC, Louder MK, O'Dell S, Schmidt SD, Phung E, Chang LA, Yap C, Todd JM, Pessaint L, Van Ry A, Browne S, Greenhouse J, Putman-Taylor T, Strasbaugh A, Campbell TA, Cook A, Dodson A, Steingrebe K, Shi W, Zhang Y, Abiona OM, Wang L, Pegu A, Yang ES, Leung K, Zhou T, Teng IT, Widge A, Gordon I, Novik L, Gillespie RA, Loomis RJ, Moliva JI, Stewart-Jones G, Himansu S, Kong WP, Nason MC, Morabito KM, Ruckwardt TJ, Ledgerwood JE, Gaudinski MR, Kwong PD, Mascola JR, Carfi A, Lewis MG, Baric RS, McDermott A, Moore IN, Sullivan NJ, Roederer M, Seder RA, Graham BS. Evaluation of the mRNA-1273 Vaccine against SARS-CoV-2 in Nonhuman Primates. N Engl J Med. 2020 Oct 15;383(16):1544-1555. doi: 10.1056/NEJMoa2024671. Epub 2020 Jul 28. PMID 32722908
- [Background] Walsh EE, Frenck RW Jr, Falsey AR, Kitchin N, Absalon J, Gurtman A, Lockhart S, Neuzil K, Mulligan MJ, Bailey R, Swanson KA, Li P, Koury K, Kalina W, Cooper D, Fontes-Garfias C, Shi PY, Tureci O, Tompkins KR, Lyke KE, Raabe V, Dormitzer PR, Jansen KU, Sahin U, Gruber WC. Safety and Immunogenicity of Two RNA-Based Covid-19 Vaccine Candidates. N Engl J Med. 2020 Dec 17;383(25):2439-2450. doi: 10.1056/NEJMoa2027906. Epub 2020 Oct 14. PMID 33053279
- [Background] Mercado NB, Zahn R, Wegmann F, Loos C, Chandrashekar A, Yu J, Liu J, Peter L, McMahan K, Tostanoski LH, He X, Martinez DR, Rutten L, Bos R, van Manen D, Vellinga J, Custers J, Langedijk JP, Kwaks T, Bakkers MJG, Zuijdgeest D, Rosendahl Huber SK, Atyeo C, Fischinger S, Burke JS, Feldman J, Hauser BM, Caradonna TM, Bondzie EA, Dagotto G, Gebre MS, Hoffman E, Jacob-Dolan C, Kirilova M, Li Z, Lin Z, Mahrokhian SH, Maxfield LF, Nampanya F, Nityanandam R, Nkolola JP, Patel S, Ventura JD, Verrington K, Wan H, Pessaint L, Van Ry A, Blade K, Strasbaugh A, Cabus M, Brown R, Cook A, Zouantchangadou S, Teow E, Andersen H, Lewis MG, Cai Y, Chen B, Schmidt AG, Reeves RK, Baric RS, Lauffenburger DA, Alter G, Stoffels P, Mammen M, Van Hoof J, Schuitemaker H, Barouch DH. Single-shot Ad26 vaccine protects against SARS-CoV-2 in rhesus macaques. Nature. 2020 Oct;586(7830):583-588. doi: 10.1038/s41586-020-2607-z. Epub 2020 Jul 30. PMID 32731257
- [Background] Wajnberg A, Amanat F, Firpo A, Altman DR, Bailey MJ, Mansour M, McMahon M, Meade P, Mendu DR, Muellers K, Stadlbauer D, Stone K, Strohmeier S, Simon V, Aberg J, Reich DL, Krammer F, Cordon-Cardo C. Robust neutralizing antibodies to SARS-CoV-2 infection persist for months. Science. 2020 Dec 4;370(6521):1227-1230. doi: 10.1126/science.abd7728. Epub 2020 Oct 28. PMID 33115920
- [Background] Chen X, Pan Z, Yue S, Yu F, Zhang J, Yang Y, Li R, Liu B, Yang X, Gao L, Li Z, Lin Y, Huang Q, Xu L, Tang J, Hu L, Zhao J, Liu P, Zhang G, Chen Y, Deng K, Ye L. Disease severity dictates SARS-CoV-2-specific neutralizing antibody responses in COVID-19. Signal Transduct Target Ther. 2020 Sep 2;5(1):180. doi: 10.1038/s41392-020-00301-9. PMID 32879307
- [Background] Hassan AO, Case JB, Winkler ES, Thackray LB, Kafai NM, Bailey AL, McCune BT, Fox JM, Chen RE, Alsoussi WB, Turner JS, Schmitz AJ, Lei T, Shrihari S, Keeler SP, Fremont DH, Greco S, McCray PB Jr, Perlman S, Holtzman MJ, Ellebedy AH, Diamond MS. A SARS-CoV-2 Infection Model in Mice Demonstrates Protection by Neutralizing Antibodies. Cell. 2020 Aug 6;182(3):744-753.e4. doi: 10.1016/j.cell.2020.06.011. Epub 2020 Jun 10. PMID 32553273
- [Background] Krammer F. SARS-CoV-2 vaccines in development. Nature. 2020 Oct;586(7830):516-527. doi: 10.1038/s41586-020-2798-3. Epub 2020 Sep 23. PMID 32967006
- [Background] 14. Muecksch F, et al. Longitudinal analysis of clinical serology assay performance and neutralising antibody levels in COVID19 convalescents. medRxiv. 2020.08.05.20169128. https://doi.org/10.1101/2020.08.05.20169128
- [Background] 15. Ripperger TJ, et al. Detection, prevalence, and duration of humoral responses to SARS-CoV-2 under conditions of limited population exposure. medRxiv. 2020.08.14.20174490; DOI: https://doi. org/10.1101/2020.08.14.20174490
- [Background] 16. Grandjean L, et al. Humoral response dynamics following infection with SARS-CoV-2. medRxiv. 2020.07.16.20155663; https://doi.org/10.1101/2020.07.16.20155663
- [Background] Iyer AS, Jones FK, Nodoushani A, Kelly M, Becker M, Slater D, Mills R, Teng E, Kamruzzaman M, Garcia-Beltran WF, Astudillo M, Yang D, Miller TE, Oliver E, Fischinger S, Atyeo C, Iafrate AJ, Calderwood SB, Lauer SA, Yu J, Li Z, Feldman J, Hauser BM, Caradonna TM, Branda JA, Turbett SE, LaRocque RC, Mellon G, Barouch DH, Schmidt AG, Azman AS, Alter G, Ryan ET, Harris JB, Charles RC. Persistence and decay of human antibody responses to the receptor binding domain of SARS-CoV-2 spike protein in COVID-19 patients. Sci Immunol. 2020 Oct 8;5(52):eabe0367. doi: 10.1126/sciimmunol.abe0367. PMID 33033172
- [Background] 18. Iyer AS. Dynamics and significance of the antibody response to SARS-CoV-2. medRxiv. 2020.07.18.20155374. DOI:10.1101/2020.07.18.20155374
- [Background] Figueiredo-Campos P, Blankenhaus B, Mota C, Gomes A, Serrano M, Ariotti S, Costa C, Nunes-Cabaco H, Mendes AM, Gaspar P, Pereira-Santos MC, Rodrigues F, Condeco J, Escoval MA, Santos M, Ramirez M, Melo-Cristino J, Simas JP, Vasconcelos E, Afonso A, Veldhoen M. Seroprevalence of anti-SARS-CoV-2 antibodies in COVID-19 patients and healthy volunteers up to 6 months post disease onset. Eur J Immunol. 2020 Dec;50(12):2025-2040. doi: 10.1002/eji.202048970. Epub 2020 Nov 10. PMID 33084029
- [Background] Isho B, Abe KT, Zuo M, Jamal AJ, Rathod B, Wang JH, Li Z, Chao G, Rojas OL, Bang YM, Pu A, Christie-Holmes N, Gervais C, Ceccarelli D, Samavarchi-Tehrani P, Guvenc F, Budylowski P, Li A, Paterson A, Yue FY, Marin LM, Caldwell L, Wrana JL, Colwill K, Sicheri F, Mubareka S, Gray-Owen SD, Drews SJ, Siqueira WL, Barrios-Rodiles M, Ostrowski M, Rini JM, Durocher Y, McGeer AJ, Gommerman JL, Gingras AC. Persistence of serum and saliva antibody responses to SARS-CoV-2 spike antigens in COVID-19 patients. Sci Immunol. 2020 Oct 8;5(52):eabe5511. doi: 10.1126/sciimmunol.abe5511. PMID 33033173
- [Background] Poland GA, Ovsyannikova IG, Kennedy RB. SARS-CoV-2 immunity: review and applications to phase 3 vaccine candidates. Lancet. 2020 Nov 14;396(10262):1595-1606. doi: 10.1016/S0140-6736(20)32137-1. Epub 2020 Oct 13. PMID 33065034
- [Background] Xia S, Duan K, Zhang Y, Zhao D, Zhang H, Xie Z, Li X, Peng C, Zhang Y, Zhang W, Yang Y, Chen W, Gao X, You W, Wang X, Wang Z, Shi Z, Wang Y, Yang X, Zhang L, Huang L, Wang Q, Lu J, Yang Y, Guo J, Zhou W, Wan X, Wu C, Wang W, Huang S, Du J, Meng Z, Pan A, Yuan Z, Shen S, Guo W, Yang X. Effect of an Inactivated Vaccine Against SARS-CoV-2 on Safety and Immunogenicity Outcomes: Interim Analysis of 2 Randomized Clinical Trials. JAMA. 2020 Sep 8;324(10):951-960. doi: 10.1001/jama.2020.15543. PMID 32789505
- [Background] Folegatti PM, Ewer KJ, Aley PK, Angus B, Becker S, Belij-Rammerstorfer S, Bellamy D, Bibi S, Bittaye M, Clutterbuck EA, Dold C, Faust SN, Finn A, Flaxman AL, Hallis B, Heath P, Jenkin D, Lazarus R, Makinson R, Minassian AM, Pollock KM, Ramasamy M, Robinson H, Snape M, Tarrant R, Voysey M, Green C, Douglas AD, Hill AVS, Lambe T, Gilbert SC, Pollard AJ; Oxford COVID Vaccine Trial Group. Safety and immunogenicity of the ChAdOx1 nCoV-19 vaccine against SARS-CoV-2: a preliminary report of a phase 1/2, single-blind, randomised controlled trial. Lancet. 2020 Aug 15;396(10249):467-478. doi: 10.1016/S0140-6736(20)31604-4. Epub 2020 Jul 20. PMID 32702298
- [Background] Zhu FC, Li YH, Guan XH, Hou LH, Wang WJ, Li JX, Wu SP, Wang BS, Wang Z, Wang L, Jia SY, Jiang HD, Wang L, Jiang T, Hu Y, Gou JB, Xu SB, Xu JJ, Wang XW, Wang W, Chen W. Safety, tolerability, and immunogenicity of a recombinant adenovirus type-5 vectored COVID-19 vaccine: a dose-escalation, open-label, non-randomised, first-in-human trial. Lancet. 2020 Jun 13;395(10240):1845-1854. doi: 10.1016/S0140-6736(20)31208-3. Epub 2020 May 22. PMID 32450106
- [Background] Zhu FC, Guan XH, Li YH, Huang JY, Jiang T, Hou LH, Li JX, Yang BF, Wang L, Wang WJ, Wu SP, Wang Z, Wu XH, Xu JJ, Zhang Z, Jia SY, Wang BS, Hu Y, Liu JJ, Zhang J, Qian XA, Li Q, Pan HX, Jiang HD, Deng P, Gou JB, Wang XW, Wang XH, Chen W. Immunogenicity and safety of a recombinant adenovirus type-5-vectored COVID-19 vaccine in healthy adults aged 18 years or older: a randomised, double-blind, placebo-controlled, phase 2 trial. Lancet. 2020 Aug 15;396(10249):479-488. doi: 10.1016/S0140-6736(20)31605-6. Epub 2020 Jul 20. PMID 32702299
- [Background] Logunov DY, Dolzhikova IV, Zubkova OV, Tukhvatullin AI, Shcheblyakov DV, Dzharullaeva AS, Grousova DM, Erokhova AS, Kovyrshina AV, Botikov AG, Izhaeva FM, Popova O, Ozharovskaya TA, Esmagambetov IB, Favorskaya IA, Zrelkin DI, Voronina DV, Shcherbinin DN, Semikhin AS, Simakova YV, Tokarskaya EA, Lubenets NL, Egorova DA, Shmarov MM, Nikitenko NA, Morozova LF, Smolyarchuk EA, Kryukov EV, Babira VF, Borisevich SV, Naroditsky BS, Gintsburg AL. Safety and immunogenicity of an rAd26 and rAd5 vector-based heterologous prime-boost COVID-19 vaccine in two formulations: two open, non-randomised phase 1/2 studies from Russia. Lancet. 2020 Sep 26;396(10255):887-897. doi: 10.1016/S0140-6736(20)31866-3. Epub 2020 Sep 4. PMID 32896291
- [Background] Jackson LA, Anderson EJ, Rouphael NG, Roberts PC, Makhene M, Coler RN, McCullough MP, Chappell JD, Denison MR, Stevens LJ, Pruijssers AJ, McDermott A, Flach B, Doria-Rose NA, Corbett KS, Morabito KM, O'Dell S, Schmidt SD, Swanson PA 2nd, Padilla M, Mascola JR, Neuzil KM, Bennett H, Sun W, Peters E, Makowski M, Albert J, Cross K, Buchanan W, Pikaart-Tautges R, Ledgerwood JE, Graham BS, Beigel JH; mRNA-1273 Study Group. An mRNA Vaccine against SARS-CoV-2 - Preliminary Report. N Engl J Med. 2020 Nov 12;383(20):1920-1931. doi: 10.1056/NEJMoa2022483. Epub 2020 Jul 14. PMID 32663912
- [Background] 28. Keech C, et al. Phase 1-2 trial of a SARS-CoV-2 recombinant spike protein nanoparticle vaccine. DOI:10.1056/NEJMoa2026920 29. 49. Zhang, Y.J. et al. Immunogenicity and safety of a SARS-CoV-2 inactivated vaccine in healthy adults aged 18-59 years: report of the randomized, double-blind, and placebo-controlled phase 2 clinical trial. medRxiv. 2020.07.31.20161216; https://doi.org/10.1101/2020.07.31.20161216
- [Background] Hotez PJ, Corry DB, Strych U, Bottazzi ME. COVID-19 vaccines: neutralizing antibodies and the alum advantage. Nat Rev Immunol. 2020 Jul;20(7):399-400. doi: 10.1038/s41577-020-0358-6. PMID 32499636
- [Background] Dagotto G, Yu J, Barouch DH. Approaches and Challenges in SARS-CoV-2 Vaccine Development. Cell Host Microbe. 2020 Sep 9;28(3):364-370. doi: 10.1016/j.chom.2020.08.002. Epub 2020 Aug 10. PMID 32798444
- [Background] Yu J, Tostanoski LH, Peter L, Mercado NB, McMahan K, Mahrokhian SH, Nkolola JP, Liu J, Li Z, Chandrashekar A, Martinez DR, Loos C, Atyeo C, Fischinger S, Burke JS, Slein MD, Chen Y, Zuiani A, Lelis FJN, Travers M, Habibi S, Pessaint L, Van Ry A, Blade K, Brown R, Cook A, Finneyfrock B, Dodson A, Teow E, Velasco J, Zahn R, Wegmann F, Bondzie EA, Dagotto G, Gebre MS, He X, Jacob-Dolan C, Kirilova M, Kordana N, Lin Z, Maxfield LF, Nampanya F, Nityanandam R, Ventura JD, Wan H, Cai Y, Chen B, Schmidt AG, Wesemann DR, Baric RS, Alter G, Andersen H, Lewis MG, Barouch DH. DNA vaccine protection against SARS-CoV-2 in rhesus macaques. Science. 2020 Aug 14;369(6505):806-811. doi: 10.1126/science.abc6284. Epub 2020 May 20. PMID 32434945
- [Background] Gao Q, Bao L, Mao H, Wang L, Xu K, Yang M, Li Y, Zhu L, Wang N, Lv Z, Gao H, Ge X, Kan B, Hu Y, Liu J, Cai F, Jiang D, Yin Y, Qin C, Li J, Gong X, Lou X, Shi W, Wu D, Zhang H, Zhu L, Deng W, Li Y, Lu J, Li C, Wang X, Yin W, Zhang Y, Qin C. Development of an inactivated vaccine candidate for SARS-CoV-2. Science. 2020 Jul 3;369(6499):77-81. doi: 10.1126/science.abc1932. Epub 2020 May 6. PMID 32376603
- [Background] Mulligan MJ, Lyke KE, Kitchin N, Absalon J, Gurtman A, Lockhart S, Neuzil K, Raabe V, Bailey R, Swanson KA, Li P, Koury K, Kalina W, Cooper D, Fontes-Garfias C, Shi PY, Tureci O, Tompkins KR, Walsh EE, Frenck R, Falsey AR, Dormitzer PR, Gruber WC, Sahin U, Jansen KU. Phase I/II study of COVID-19 RNA vaccine BNT162b1 in adults. Nature. 2020 Oct;586(7830):589-593. doi: 10.1038/s41586-020-2639-4. Epub 2020 Aug 12. PMID 32785213
- [Background] Sahin U, Muik A, Derhovanessian E, Vogler I, Kranz LM, Vormehr M, Baum A, Pascal K, Quandt J, Maurus D, Brachtendorf S, Lorks V, Sikorski J, Hilker R, Becker D, Eller AK, Grutzner J, Boesler C, Rosenbaum C, Kuhnle MC, Luxemburger U, Kemmer-Bruck A, Langer D, Bexon M, Bolte S, Kariko K, Palanche T, Fischer B, Schultz A, Shi PY, Fontes-Garfias C, Perez JL, Swanson KA, Loschko J, Scully IL, Cutler M, Kalina W, Kyratsous CA, Cooper D, Dormitzer PR, Jansen KU, Tureci O. COVID-19 vaccine BNT162b1 elicits human antibody and TH1 T cell responses. Nature. 2020 Oct;586(7830):594-599. doi: 10.1038/s41586-020-2814-7. Epub 2020 Sep 30. PMID 32998157
- [Background] Bos R, Rutten L, van der Lubbe JEM, Bakkers MJG, Hardenberg G, Wegmann F, Zuijdgeest D, de Wilde AH, Koornneef A, Verwilligen A, van Manen D, Kwaks T, Vogels R, Dalebout TJ, Myeni SK, Kikkert M, Snijder EJ, Li Z, Barouch DH, Vellinga J, Langedijk JPM, Zahn RC, Custers J, Schuitemaker H. Ad26 vector-based COVID-19 vaccine encoding a prefusion-stabilized SARS-CoV-2 Spike immunogen induces potent humoral and cellular immune responses. NPJ Vaccines. 2020 Sep 28;5:91. doi: 10.1038/s41541-020-00243-x. eCollection 2020. PMID 33083026
- [Background] Bubar KM, Reinholt K, Kissler SM, Lipsitch M, Cobey S, Grad YH, Larremore DB. Model-informed COVID-19 vaccine prioritization strategies by age and serostatus. Science. 2021 Feb 26;371(6532):916-921. doi: 10.1126/science.abe6959. Epub 2021 Jan 21. PMID 33479118
- [Background] Gaebler C, Nussenzweig MC. All eyes on a hurdle race for a SARS-CoV-2 vaccine. Nature. 2020 Oct;586(7830):501-502. doi: 10.1038/d41586-020-02926-w. No abstract available. PMID 33077943
- [Background] Trabaud MA, Icard V, Milon MP, Bal A, Lina B, Escuret V. Comparison of eight commercial, high-throughput, automated or ELISA assays detecting SARS-CoV-2 IgG or total antibody. J Clin Virol. 2020 Nov;132:104613. doi: 10.1016/j.jcv.2020.104613. Epub 2020 Sep 7. PMID 32942137
- [Background] Houlihan CF, Beale R. The complexities of SARS-CoV-2 serology. Lancet Infect Dis. 2020 Dec;20(12):1350-1351. doi: 10.1016/S1473-3099(20)30699-X. Epub 2020 Sep 23. No abstract available. PMID 32979317
- [Background] National SARS-CoV-2 Serology Assay Evaluation Group. Performance characteristics of five immunoassays for SARS-CoV-2: a head-to-head benchmark comparison. Lancet Infect Dis. 2020 Dec;20(12):1390-1400. doi: 10.1016/S1473-3099(20)30634-4. Epub 2020 Sep 23. PMID 32979318
- [Background] Rosadas C, Randell P, Khan M, McClure MO, Tedder RS. Testing for responses to the wrong SARS-CoV-2 antigen? Lancet. 2020 Sep 5;396(10252):e23. doi: 10.1016/S0140-6736(20)31830-4. Epub 2020 Aug 28. No abstract available. PMID 32866429
- [Background] Long QX, Tang XJ, Shi QL, Li Q, Deng HJ, Yuan J, Hu JL, Xu W, Zhang Y, Lv FJ, Su K, Zhang F, Gong J, Wu B, Liu XM, Li JJ, Qiu JF, Chen J, Huang AL. Clinical and immunological assessment of asymptomatic SARS-CoV-2 infections. Nat Med. 2020 Aug;26(8):1200-1204. doi: 10.1038/s41591-020-0965-6. Epub 2020 Jun 18. PMID 32555424
- [Background] Seow J, Graham C, Merrick B, Acors S, Pickering S, Steel KJA, Hemmings O, O'Byrne A, Kouphou N, Galao RP, Betancor G, Wilson HD, Signell AW, Winstone H, Kerridge C, Huettner I, Jimenez-Guardeno JM, Lista MJ, Temperton N, Snell LB, Bisnauthsing K, Moore A, Green A, Martinez L, Stokes B, Honey J, Izquierdo-Barras A, Arbane G, Patel A, Tan MKI, O'Connell L, O'Hara G, MacMahon E, Douthwaite S, Nebbia G, Batra R, Martinez-Nunez R, Shankar-Hari M, Edgeworth JD, Neil SJD, Malim MH, Doores KJ. Longitudinal observation and decline of neutralizing antibody responses in the three months following SARS-CoV-2 infection in humans. Nat Microbiol. 2020 Dec;5(12):1598-1607. doi: 10.1038/s41564-020-00813-8. Epub 2020 Oct 26. PMID 33106674
- [Background] Ibarrondo FJ, Fulcher JA, Goodman-Meza D, Elliott J, Hofmann C, Hausner MA, Ferbas KG, Tobin NH, Aldrovandi GM, Yang OO. Rapid Decay of Anti-SARS-CoV-2 Antibodies in Persons with Mild Covid-19. N Engl J Med. 2020 Sep 10;383(11):1085-1087. doi: 10.1056/NEJMc2025179. Epub 2020 Jul 21. No abstract available. PMID 32706954
- [Background] 45. https://www.siemens-healthineers.com/en-us/laboratory-diagnostics/assays-by-diseases-conditions/infectious-disease-assays/sars-cov-2-igg-assay